CLINICAL TRIAL: NCT04204512
Title: Comparison of 2 Probes Frequencies in the Diagnosis of Giant Cell Arteritis
Brief Title: Comparison of 22Mhz and 18Mhz High-frequency Probes for the Ultrasound Study of Temporal Arteries in Patients Suspected of Having Giant Cell Arteritis
Acronym: ECHORTON
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ECHORTON (29BRC19.0275)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Giant Cell Arteritis
Keywords: ultrasound,; giant cell arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the structural features of temporal arteritis using two frequencies probes: 18 and 22Mhz.

DETAILED DESCRIPTION:
Comparison of the results obtained by using 2 different frequencies probes in the diagnosis of giant cell arteritis

ELIGIBILITY:
Inclusion Criteria:

* sedimentation rate> 50 mm/h or recent unusual headache or unusual fever, recent visual trouble or jaw claudication, or induration temporal arteritis

Exclusion Criteria:

* previous diagnosis of giant cell arteritis and relapse of the giant cell arteritis and opposition to participate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspicion of giant cell arteritis
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
halo sign of temporal arteritis | inclusion
  hypoechogenicity of the wall artery
compression sign of of temporal arteritis | inclusion
  persistent of increased inflammatory arteries wall

SECONDARY OUTCOMES:
halo sign of carotid arteritis | inclusion
  hypoechogenicity of the wall artery
halo sign of subclavian arteritis | inclusion
  hypoechogenicity of the wall artery
halo sign of axillary arteritis | inclusion
  hypoechogenicity of the wall artery
other structural abnormalities in unilateral B mode | inclusion
  stenosis, occlusion
other structural abnormalities in bilateral B mode | inclusion
  stenosis, occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 18 month and ending five years following the end of study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.